CLINICAL TRIAL: NCT02315326
Title: A Phase I/II Trial of the Bruton's Tyrosine Kinase (BTK) Inhibitor, Ibrutinib, in Patients With Newly Diagnosed or Refractory/Recurrent Primary Central Nervous System Lymphoma (PCNSL) and Refractory/Recurrent Secondary Central Nervous System Lymphoma (SCNSL)
Brief Title: Bruton's Tyrosine Kinase (BTK) Inhibitor, Ibrutinib, in Patients With Newly Diagnosed or Refractory/Recurrent Primary Central Nervous System Lymphoma (PCNSL) and Refractory/Recurrent Secondary Central Nervous System Lymphoma (SCNSL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Pharmacyclics LLC. (Industry); Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 14-184
Record Dates: First submitted 2014-12-09; First posted 2014-12-11 (Estimated); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Adult Patients With Newly Diagnosed or Relapsed or Refractory Primary Central Nervous System Lymphoma (PCNSL); Or Relapsed or Refractory Secondary Central Nervous System Lymphoma (SCNSL)
Keywords: Ibrutinib,; Imbruvica™; Bruton's Tyrosine Kinase (BTK) Inhibitor; HD-MTX; 14-184
MeSH Terms: conditions — Recurrence | interventions — ibrutinib; Rituximab; Procarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: Participants with refractory/recurrent PCNSL or refractory/recurrent SCNSL (Experimental): This is an open-label, non-randomized, single center, dose escalation, phase I/II study to establish the maximum-tolerated dose (MTD) of ibrutinib as a single agent in patients with refractory/recurrent PCNSL or refractory/recurrent SCNSL (Arm A).
  Interventions: Drug: Ibrutinib; Drug: HD- Methotrexate (MTX); Drug: Rituximab + HD- Methotrexate (MTX)
- Arm B: Participants with refractory/recurrent PCNSL or refractory/recurrent SCNSL (Experimental): The defined MTD from Arm A will then be used in an expansion cohort to further assess toxicity and clinical activity
  Interventions: Drug: Ibrutinib; Drug: HD- Methotrexate (MTX); Drug: Rituximab + HD- Methotrexate (MTX)
- Arm C: Participants with refractory/recurrent PCNSL or refractory/recurrent SCNSL (Experimental): Arm C will investigate the MTD of ibrutinib in combination with HD-MTX and to determine the safety and tolerability of the ibrutinib/HD-MTX combination regimen in PCNSL and SCNSL patients. To minimize drug-drug interaction between HD-MTX and Ibrutinib, Ibrutinib will not be administered concurrently with HD-MTX.
  Interventions: Drug: Ibrutinib; Drug: HD- Methotrexate (MTX); Drug: Rituximab + HD- Methotrexate (MTX)
- Arm D: Participants with refractory/recurrent PCNSL or refractory/recurrent SCNSL (Experimental): THIS IS ONLY ARM RECRUITING In Arm D, patients will be treated with 4 cycles of therapy. Methotrexate (3.5 g/m2) will be given at Dday 1 and Dday 15 of each cycle. Rituximab (500 mg/m2) will be given at Dday 0 and Dday 15 of each cycle. Vincristine (1.4mg/m2) will be given at Dday 1 and 15 of cycle 1 and 2 only. Procarbazine (100mg/m2) will be given of Day 1 of each cycle. Ibrutinib will be dosed at 560 mg daily. Arm D will have a safety lead-in of 6 patients. If more than 1 of 6 subjects develop a dose limiting toxicity (DLT) within the first 28 days of therapy (cycle 1), ibrutinib will be reduced to 420 mg daily dosing, and 6 additional patients will be enrolled. If more than 1 of 6 subjects develop a DLT, additional enrollment will be stopped.
  Interventions: Drug: Ibrutinib; Drug: HD- Methotrexate (MTX); Drug: Rituximab + HD- Methotrexate (MTX); Drug: procarbazine

INTERVENTIONS:
Drug: Ibrutinib — Arm A: Ibrutinib will be given once daily. The starting dose cohort (level 1) will receive 560 mg/day (4 x 140 mg capsules). During the dose escalation period of the study, the "3+3" design will be applied (see Table 3). Participants will be assigned to cohorts of increasing oral daily doses of ibrutinib (560mg, 840mg) until disease progression, intolerable toxicity or death. Three patients with recurrent/refractory PCNSL or recurrent/refractory SCNSL will be treated with daily oral ibrutinib for a 28-day cycle starting at dose level 1 and observed for toxicities during cycle 1. Arm B: Ibrutinib will be given at the MTD defined in Arm A.
  Other Names: Imbruvica™
Drug: HD- Methotrexate (MTX) — Arm C1: HD-MTX at 3.5g/m2 (standard hydration/leucovorin support) will be given on day 1 and 15 of each 28-day cycle for a total of 4 cycles totaling 8 HD-MTX administrations. Ibrutinib will be given between days 5 and 14 as well as days 19 and 28 of each cycle and continued daily after completion of HD-MTX treatments.The starting dose of ibrutinib is 560 mg/day (4x140mg capsules)
Drug: Rituximab + HD- Methotrexate (MTX) — Arm C2: Intravenous rituximab (500mg/m2) will be given on day 0, 14, and 28 of cycle 1 and day 14 and 28 of all following cycles. HD-MTX at 3.5g/m2 (standard hydration/leucovorin support) will be given on day 1 and 15 of each 28-day cycle for a maximum of 4 cycles totaling 8 HD-MTX administrations. Ibrutinib will be given between days 5 and 14 as well as days 19 and 28 of each cycle and continued daily after completion of HD-MTX treatments. The starting dose of ibrutinib is 560 mg/day (4x140mg capsules; dose level 1) (see Table 4). Filgrastim will be given at days 7-11 and 22-26.
Drug: procarbazine — Arm D: THIS IS THE ONLY ARM RECRUITING: : Oral procarbazine (100mg/m2/day) will be given on Day 1 through 7 during each cycle. Patients will be maintained on a tyramine-free diet during procarbazine administration.
  Arms: Arm D: Participants with refractory/recurrent PCNSL or refractory/recurrent SCNSL

SUMMARY:
The purpose of this study is to test any good or bad effects of the study drug called of ibrutinib (also known as Imbruvica™). At this stage of this trial, the study is investigating whether Ibrutinib can be incorporated into the established first-line chemotherapy regimen rituximab, methotrexate, vincristine, and procarbazine (R-VMP) in order to further refine the first-line induction therapy for PCNSL, as observed by a superior CRR (complete response rate) (ARM D RECRUITING ONLY)

ELIGIBILITY:
The population consists of adult patients with newly diagnosed or relapsed or refractory primary central nervous system lymphoma (PCNSL) or relapsed or refractory secondary central nervous system lymphoma (SCNSL)

Patients eligible for inclusion in this study have to meet all the following criteria:

Inclusion Criteria:

* Participants must be able to understand and be willing to sign a written informed consent document
* Men and woman who are at least 18 years of age on the day of consenting to the study
* Histologically or cystologically documented PCNSL or histologically documented systemic diffuse large B-cell lymphoma (DLBCL)
* Patients must have relapsed/refractory PCNSL or relapsed/refractory SCNSL (Arm A, B, C) or newly diagnosed PCNSL (Arm D)
* All patients need to have received at least one prior CNS directed therapy. There is no restriction on the number of recurrences (Arm A, B , C only)
* Patients with parenchymal lesions must have unequivocal evidence of disease progression on imaging (MRI of the brain or head CT) 21 days prior to study registration. For patients with leptomeningeal disease only, CSF cytology must document lymphoma cells and/or imaging findings consistent with CSF disease 21 days prior to study registration (at the discretion of the investigator) (Arm A, B , C only).
* Participants must have an ECOG performance status of 0, 1, or 2
* Within the past 21 days prior to study registration (for Arm D: prior to treatment initiation) participants must have adequate bone marrow and organ function shown by:

  * Absolute neutrophil count (ANC) ≥ 0.75 x 109/L
  * Platelets ≥ 75 x 109/L and no platelet transfusion within the past 21 days prior to study registration
  * Hemoglobin (Hgb) ≥ 8 g/dL and no red blood cell (RBC) transfusion within the past 21 days prior to study registration
  * International Normalized Ratio (INR) ≤ 1.5 and PTT (aPTT) ≤ 1.5 times the upper limit of normal
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the upper limit of normal
  * Serum bilirubin ≤ 1.5 times the upper limit of normal; or total bilirubin ≤ 3 times the upper limit of normal with direct bilirubin within the normal range in patients with well documented Gilbert Syndrome
  * Serum creatinine ≤ 2 times the upper limit of normal
  * Arm C: calculated creatinine clearance(CrCl) > 50ml/min using the Cockcroft-Gault equation (Men: CrCl (min/ml) = (140-age) X (actual weight in kg) / 72 X serum creatinine (mg/dL); Women: CrCl (ml/min) = (140-age) X (actual weight in kg) X 0.85 / 72 X serum creatinine (mg/dL))
* Woman of reproductive potential must agree to use highly effective methods of birth control during the period of therapy and for 30 days after the last dose of the study drug. Men who are sexually active must agree to use highly effective contraception during the period of therapy and for 3 months after the last dose
* Female subjects of childbearing potential must have a negative plasma pregnancy test upon study entry. See section on Pregnancy and Reproduction
* Patients must be able to tolerate MRI/CT scans
* Patients must be able to tolerate lumbar puncture and/or Ommaya taps
* Participants must have recovered to grade 1 toxicity from prior therapy (Arm A, B , C only)
* Participates must be able to submit 20 unstained formalin-fixed, paraffin-embedded (FFPE) slides from the initial tissue diagnosis prior to study registration for confirmation of diagnosis and correlative studies Arm C1 and C2: SCNSL patients do not require one prior CNS directed treatment. Newly diagnosed SCNSL patients are eligible as long as their systemic disease has been treated and does not require any active treatment.

Arm D: PCNSL patients without one prior CNS directed treatment.

Exclusion Criteria:

* Patients with SCNSL actively receiving treatment for extra-CNS disease are excluded
* Patient is concurrently using other approved or investigational antineoplastic agents. Investigational supportive agents are permitted.
* Patient has received chemotherapy, monoclonal antibodies or targeted anticancer therapy ≤ 4 weeks or 5 half-lives, whichever is shorter, or 6 weeks for nitrosurea, or mitomycin-C prior to starting the study drug, or the patient has not recovered from the side effects of such therapy Patient has received external beam radiation therapy to the CNSwithin 21 days of the first dose of the study drug
* Patient requires more than 8 mg of dexamethasone daily or the equivalent therapy (Arm A, B , C only)
* Patient has an active concurrent malignancy requiring active therapy
* The patient has been treated with radio- or toxin-immunoconjugates within 70 days of the first dose of the study drug
* Patient has previously taken is allergic to components of the study drug. For Arms A and B only: Patient has previously taken ibrutinib.
* Patient is using warfarin or any other Coumadin-derivative anticoagulant or vitamin K antagonists. Patients must be off warfarin-derivative anticoagulants for at least seven days prior to starting the study drug. Low molecular weight heparin is allowed. Patients with congenital bleeding diathesis are excluded
* Patient is taking a drug known to be a moderate and strong inhibitor or inducers of the P450 isoenzyme CYP3A. Participants must be off P450/CYP3A inhibitors and inducers for at least two weeks prior to starting the study drug
* Patient is using systemic immunosuppressant therapy, including cyclosporine A, tacrolimus, sirolimus, and other such medications, or chronic administration of > 5 mg/day or prednisone or the equivalent. Participants must be off of immunosuppressant therapy for at least 28 days prior to the first dose of the study drug
* Patient has significant abnormalities on screening electrocardiogram (EKG) and active and significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, hypertension, valvular disease, pericarditis, or myocardial infarction within 6 months of screening
* Patient has a known bleeding diathesis (e.g. von Willebrand's disease) or hemophilia
* Patient is known to have human immunodeficiency virus (HIV) infection
* Patient is known to have a history of active or chronic infection with hepatitis C virus (HCV) or hepatitis B virus (HBV) as determined by serologic tests
* Patient is known to have an uncontrolled active systemic infection
* Patient underwent major systemic surgery ≤ 2 weeks prior to starting the trial treatment or who has not recovered from the side effects of such surgery, or who plan to have surgery within 2 weeks of the first dose of the study drug therapy (Arm A, B , C only).
* Patient is unable to swallow capsules or has a disease or condition significantly affecting gastrointestinal function, such as malabsorption syndrome, resection of the stomach or small bowel, or complete bowel obstruction
* Patient has poorly controlled diabetes mellitus with a glycosylated hemoglobin >8% or poorly controlled steroid-induced diabetes mellitus with a glycosylated hemoglobin of >8%
* Patient has a life-threatening illness, medical condition, or organ system dysfunction that, in the opinion of the investigator, could compromise the subject's safety or put the study outcomes at undue risk
* Women who are pregnant or nursing (lactating), where pregnancy is defined as a state of a female after conception until the termination of gestation, confirmed by a positive serum hCG laboratory test of > 5 mIU/mL (See section on Pregnancy and Reproduction)
* Patient has undergone prior allogenic stem cell transplant (autologous stem cell transplant is NOT an exclusion)
* The patient is unwell or unable to participate in all required study evaluations and procedures
* Patient is unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations. A legal representative can consent on behalf of a patient who is able to understand the purpose and risk of the study but not able to provide a signature on the ICF and authorization to use PHI due to neurologic deficits (e.g. motor or language deficits) (Arm A, B , C only)

Arm C and D: Patients with a methotrexate allergies are excluded.

Arm D: Patients with pre-existing peripheral motor or sensory neuropathy ≥ grade 3 (CTCAE 5.0)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2014-12-08 (Actual); Primary Completion 2026-01-28 (Actual); Study Completion 2026-01-28 (Actual)

PRIMARY OUTCOMES:
define the Maximum Tolerated Dose (MTD) of ibrutinib (phase I) | 1 year
  A standard 3+3 design will be employed. Three dose levels of ibrutinib will be investigated. Patients will be treated in cohorts of size three to six and the dosage will be escalated if the clinical toxicity is acceptable. A dose-limiting toxicity (DLT) is defined as in any of the following during cycle 1: any grade 4 hematologic toxicity, grade 3 febrile neutropenia and grade 3 thrombocytopenia associated with bleeding or any grade 3 non-hematologic toxicity that does not respond to supportive therapy and at least possibly related to treatment with ibrutinib.
progression free survival (phase II) | 2 years
  Progression-free survival (PFS) is defined as the time from the date of treatment start to the date of the first documented PD or death due to any cause.
define the Maximum Tolerated Dose (MTD) of ibrutinib in combination with high-dose Methotrexate (HD-MTX) | 1 year
  Three patients with PCNSL or SCNSL will be treated with daily oral ibrutinib +/- HD-MTX for a 28-day cycle starting at dose level 1 and observed for toxicities for a minimum of 4 weeks. Dose-limiting toxicity (DLT) will be defined as any grade 4 hematologic toxicity, grade 3 febrile neutropenia and grade 3 thrombocytopenia associated with bleeding as well as any grade 3 non-hematologic toxicity that does not respond to supportive therapy and at least possibly related to ibrutinib. If no DLT is observed in any of the 3 treated patients, we will escalate to the next dose level.

SECONDARY OUTCOMES:
safety/tolerability of ibrutinib in patients by assessing the frequency and severity of adverse events | 1 year
  in patients by assessing the frequency and severity of adverse events.
  1. The severity grade (CTCAE Grade 1-4)
  2. Its duration (Start and end dates)
  3. Its relationship to the study treatment (Reasonable possibility that AE is related: No, Yes)
  4. Action taken with respect to study or investigational treatment (none, dose adjusted, temporarily interrupted, permanently discontinued, unknown, ongoing, not applicable)
progression free survival | 16 weeks, 24 weeks & 48 weeks
  Progression-free survival (PFS) is defined as the time from the date of treatment start to the date of the first documented PD or death due to any cause.
Duration of response | 2 years
  Duration of response is defined as the time from the date of first occurrence of CR or PR to the date of the first documented PD or death due to any cause.Duration of response will be described using Kaplan-Meier curves with appropriate summary statistics

CONTACTS AND LOCATIONS:
Overall Officials: Christian Grommes, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

REFERENCES:
- [Derived] Krebs S, Mauguen A, Yildirim O, Hatzoglou V, Francis JH, Schaff LR, Mellinghoff IK, Schoder H, Grommes C. Prognostic value of [18F]FDG PET/CT in patients with CNS lymphoma receiving ibrutinib-based therapies. Eur J Nucl Med Mol Imaging. 2021 Nov;48(12):3940-3950. doi: 10.1007/s00259-021-05386-0. Epub 2021 May 8. PMID 33966087
- [Derived] Grommes C, Tang SS, Wolfe J, Kaley TJ, Daras M, Pentsova EI, Piotrowski AF, Stone J, Lin A, Nolan CP, Manne M, Codega P, Campos C, Viale A, Thomas AA, Berger MF, Hatzoglou V, Reiner AS, Panageas KS, DeAngelis LM, Mellinghoff IK. Phase 1b trial of an ibrutinib-based combination therapy in recurrent/refractory CNS lymphoma. Blood. 2019 Jan 31;133(5):436-445. doi: 10.1182/blood-2018-09-875732. Epub 2018 Dec 19. PMID 30567753
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/